CLINICAL TRIAL: NCT04180059
Title: A Phase 1 Dose-escalation Study Testing the Feasibility and the Tolerance of Infusion of a Specific Third Party Suicide Gene-transduced Anti-HLA-DPB1*0401 CD4+ T Cell Clone in HLA-DPB1*04:01 Positive Tumor Recipients Receiving an Allotransplant From a HLA-DPB1*04:01 Negative Donor.
Brief Title: Phase I Study of CTL Anti-DP Infusion Post-hematopoietic Stem Cell Transplantation
Acronym: CTL-DP 01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC16_0157
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Haematologic Disease
Keywords: hematopoietic stem cell transplantation; lymphocyte infusion; cytotoxic T lymphocyte; HLA-DP; T cell therapy
MeSH Terms: conditions — Hematologic Diseases | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: Biological, T cell clone
  A standard phase 1 dose-escalation study will be used:
  Level 1: 1 x 10^4 cells/kg of recipient, Level 2: 5 x 10^4 cells/kg, Level 3: 25 x 10^4 cells/kg, Level 4: 50 x 10^4 cells/kg, Level 5: 100 x 10^4 cells/kg.
  After study of toxicity of the 4 injected patients, choice has been made to stop the CRM method to choose the dose and to test only 2 doses for each last patients : 100 x 10^4 cells/kg (actual level 5) and 500 x 10^4 cells/kg (choice based on compassionnal injections data at the level 5)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CTL 19 : T cell therapy (Experimental): Level 1: 1 x 104 cells/kg of recipient, Level 2: 5 x 104 cells/kg, Level 3: 25 x 104 cells/kg, Level 4: 50 x 104 cells/kg, Level 5: 100 x 104 cells/kg. After study of toxicity of the 4 injected patients, choice has been made to stop the CRM method to choose the dose and to test only 2 doses for each last patients : 100 x 10^4 cells/kg (actual level 5) and 500 x 10^4 cells/kg (choice based on compassionnal injections data at the level 5)
  Interventions: Combination Product: CTL 19

INTERVENTIONS:
Combination Product: CTL 19 — Patients candidate for allogeneic transplantation who are both HLA-DPB1*04:01 and with a HLA-DPB1*04:01-expressing hematological malignancy (almost 100% of cases) with a donor HLA-DPB1*04:01 negative, will be proposed to receive one single infusion of the T cell clone at 4-5 months post-transplantation, once the immunosuppression by cyclosporine and/or mycophenolate mofetil has been discontinued.
  Other Names: T cell therapy

SUMMARY:
For several decades, allogeneic hematopoietic stem cell trans-plantation (allo-HSCT) has remained an important strategy in the management of patients with high-risk hematological malignancies. The acceptance of umbilical cord blood (UCBT) and haploidentical grafts (Haplo) as viable alternative donors for allo-HSCT has increased the options for patients with no matched donors and now ensures that a donor can be identified for virtually all patients. Relapsed disease is a principal threat to these patients and affects 30-50% of them. The therapeutic options for these relapsing patients are diverse but remain largely ineffective in altering their long-term outcomes. Therefore, pre-emptive treatment post allo-HSCT is considered.

MHC (major histocompatibility complex) class II molecules are a family of molecules normally found only on hematopoietic cells. cell-surface proteins are responsible for the regulation of the immune system in humans and are important in disease defense.

They are the major cause of organ transplant rejections. Different HLA-DPB1 alleles exist in the general population. HLA-DPB1*04:01 is the most frequent (70.5%) while HLA-DPB1*02:01 represents 32% and HLA-DPB1*03:01 20%. In allo-HSCT, the donor and the recipient may express different HLA-DPB1 molecules. HLA-DPB1 matching status has an impact on GVL (graft versus leukemia) and GVHD. In recipients of HSCT, a match for DPB1 is associated with a significantly increased risk of disease relapse, irrespective of the matching status of other HLA molecules.. Therefore, one could anticipate that a mismatched of HLA class II could induce a selective GVL reactivity without GVHD.

HLA-DP-expressing B cell and myeloid malignancies can be recognized and lysed by HLA-DP-specific T cells. The majority of leukemic cells (Acute Myeloid Leukemia, Acute Lymphoid Leukemia, Chronic Lymphoid Leukemia) express HLA-DP. A T cell clone recognizing specifically HLA-DPB1*0401 has been developed as a permanent cell line This clone has been demonstrated to be able to kill HLA-DPB1*0401 positive leukemic cells. In addition, this clone harbors a special suicide gene allowing the destruction of the clone in presence of a specific anti-viral drug named ganciclovir.

We hypothesize that infusion of a third party suicide gene-transduced T cell clone directed against HLA-DPB1*401 might protect against possible relapse of hematological malignancies.

We propose to inject iv escalating dose of a third party clone recognizing HLA-DPB1*04:01, 4 to 5 months following transplantation (when immunosuppressive drugs have been discontinued) in patients HLA-DPB1*04:01 positive with a donor HLA-DPB1*04:01 negative to evaluate the feasibility, toxicity, benefits of this immune intervention.

DETAILED DESCRIPTION:
Rationale Despite graft-versus-tumor effect, relapse remains one of the main causes of morbidity and mortality in allo-HSCT recipients. Forty to 50% of deaths following allo-HSCT are due to disease relapse. In case of relapse, the prognosis is very poor and disease burden remains a challenge for the use of adoptive cellular therapy alone. The 3 year overall survival (OS) in case of post-transplant relapse is dismal. The post-transplant period is characterized by a prolonged phase of immunodeficiency leading to increased vulnerability to infections and risk of relapse. For this reason, maintenance or pre-emptive therapies for patients in CR (complete remission) are now considered to prevent future relapse. Following allo-HSCT, the recognition by donor T lymphocytes of recipient HLA antigens may result in different consequences. On one side, T cells may recognize antigens present on malignant cells and eradicate residual disease or prevent tumor relapse. On the other side, injection of unselected T cells may induce a graft-versus-host-disease (GVHD).

HLA-DPB1 is one of MHC class II molecule lying centromeric to other class II loci on chromosome 6p21.3. Increase recombination events are found in the region between the HLA-DP loci and other class II loci, explaining the relative lack of linkage disequilibrium (LD) between HLA-DP (* HLA- DP: Human Leucocytes Antigen (DP allele))and the rest of MHC haplotype. For this reason, it is difficult to find a donor matched for DPB1 in addition to other classic HLA molecules. In sibling donors, the rate of incompatibility has been estimated to be as high as 10.9% and in unrelated donors a mismatch rate can be up to 89%. HLA-DPB1 is often not taken into consideration in donor selection. However HLA-DPB1 matching status has an impact on GVL and GVHD. In recipients of HSCT, a match for DPB1 is associated with a significantly increased risk of disease relapse, irrespective of the matching status of other HLA molecules. HLA class II molecules expression is mainly restricted to hematopoietic cells. Therefore, one could anticipate that a mismatched of HLA class II could induce a selective GVL reactivity without GVHD. However, HLA class II expression can be upregulated on various tissues following exposure to pro-inflammatory cytokines with a risk of GVHD as it is the case following some conditioning regimens or infections.

The frequency of the different HLA-DPB1 alleles in the general population is well known: HLA-DPB1*04:01 is the most frequent (70.5%) HLA-DPB1*02:01 and and HLA-DPB1*03:01 represent 32% and 20% respectively. 96% of leukemic cells could potentially be targeted with only three CTL clones directed against HLA-DPB1*04:01, 03:01 and 02:01.

HLA-DP-expressing B cell and myeloid malignancies can be recognized and lysed by HLA-DP-specific CD4+ cells ( CD4+ : cluster of differentiation 4+). The majority of leukemic cells (AML, ALL, CLL) express HLA-DP. CD4+ cytotoxic T cell (CTL) clones recognizing specifically HLA-DPB1*04:01 can be identified and have been demonstrated to be able to kill HLA-DPB1*04:01 positive leukemic cells.

In addition, it has already been shown that HLA-DP-specific CD4+ T cells can induce graft-versus-leukemia reactivity in the presence or absence of graft-versus-host disease. In this study the presence of HLA-DP-specific CD4+ T cells correlated with the clinical response to DLI.

The team of the Inserm unit 1232 (H. Vié, B. Clemenceau, both co-investigators of this project) has developed a suicide gene-transduced CD4+ T cell clone that recognizes the HLA-DPB1*401, which is the most frequent HLA-DPB1 allele expressed by leukemic blasts (70%). This clone has been described in detailed in :"The doubling potential of T lymphocytes allows clinical-grade production of a bank of genetically modified monoclonal T-cell populations" by Vivien R et al. Cytotherapy. 2018 Mar;20(3):436-452.

Several clinical trials have evaluated the possibility to inject, following allo-HSCT, donor lymphocytes transduced with a suicide gene either to treat tumor relapse or to accelerate the immune reconstitution. No acute infusion-related toxicity has been reported. Ganciclovir was used in some patients to control GVHD, leading to a rapid elimination of TK+ cells (tyrosine kinase +).

The clone was obtained by performing a mixed lymphocytes culture (MLR) between two populations differing only by HLA-DP, and subsequently by transducing reactive T cells with high efficiency, and finally cloning them directly, before selecting each clone for the desired characteristics. Thanks to a clinical grade Herpes-simplex-virus-TK vector, the clone harbors a suicide gene and can be killed in presence of ganciclovir (GCV).

This clone presents several important characteristics in terms of efficiency and safety. The clone is stable following thawing. It can be grown and amplified in vitro following thawing (at least more than one million times), while maintaining its cytotoxic capacity. It produces TH1-type cytokines in large amounts.

Regarding the safety of the CTL antiDP under study, we emphasized on two major points: Specificity and sensitivity to ganciclovir:

Specificity. The clone is specific for HLA-DPB1*04:01. The clone was selected against a donor homozygous for HLA-DPB1*04:01 (and identical for HLA-A, B, C, DQ, DR). Specificity testing confirmed the recognition of HLA-DPB1*:04:01. Yet, HLA-DPB1 alleles described are numerous (447 proteins to date IMGT (ImMunoGeneTics database)/HLA release, www.ebi.ac.uk/ipd/index.html), and it is just impossible to anticipate the cross reactions exhaustively (beyond some against HLA-DPB1*04:02 and HLA-DPB1*05:01 that have been observed against particular cell lines). The risk, since we are in a context of allo-HSCT, would be the recognition of donor cells and thus a possibility of graft rejection. For this reason, we will perform a pre-inclusion testing where donor cells will be used as targets for the clone.

Sensitivity to ganciclovir (GCV) : The proliferation tests in the presence of GCV confirms the efficacy of GCV with sufficient margin according to GCV blood levels reached during a conventional treatment.

Data from our colleagues show a low number of T cells detectable during the first months post-transplant, with a relative increased of Treg cells meaning that the clone may not be eliminated rapidly by donor T-cells.

The reasons to administer a suicide gene-transduced CD4+ T cell clone recognizing HLA-DPB1*04:01 following allogeneic transplantation can be summarized in the following points :

1. Relapse of the hematological malignancy remains a serious concern in these types of transplantation.

3. The immune reconstitution is very delayed allowing for injection of a third party T cell clone.

4. In case of GVHD following the CTL infusion, the CTL clone can be rapidly eliminated using ganciclovir.

Hypothesis We hypothesize that the infusion of a third party suicide gene-transduced T cell clone directed against HLA-DPB1*04:01 following allogeneic transplantation can be safe and might protect against possible relapse of hematological malignancies

Detailed description of the methodology (number of necessary subjects) Patients candidate for allogeneic transplantation who are both HLA-DPB1*04:01 and with aHLA-DPB1*04:01-expressing hematological malignancy (almost 100% of cases) with a donor HLA-DPB1*04:01 negative, will be proposed to receive one single infusion of the T cell clone at 4-5 months post-transplantation, once the immunosuppression by cyclosporine and/or mycophenolate mofetil has been discontinued. The expression of HLA-DPB1* by tumor cells will be checked by cytometry or immunohistochemistry. Any possible cross-reactivity of the clone against donor cells will also be excluded

A standard phase 1 dose-escalation study will be used:

Level 1: 1 x 104 cells/kg of recipient, Level 2: 5 x 104 cells/kg, Level 3: 25 x 104 cells/kg, Level 4: 50 x 104 cells/kg, Level 5: 100 x 104 cells/kg. After study of toxicity of the 4 injected patients, choice has been made to stop the CRM method to choose the dose and to test only 2 doses for each last patients : 100 x 10^4 cells/kg (actual level 5) and 500 x 10^4 cells/kg (choice based on compassionnal injections data at the level 5). All the more, if a DLT was observed at a dose of 100.10^4 cells/kg (see definition in paragraph 2.1.2), and after advice from the DSMB, a 2nd patient would be included and injected at the same dose, to confirm that the MTD had indeed been reached.

* Should MTD be confirmed in this 2nd patient, the study would be terminated.
* In the absence of MTD in this 2nd patient, and on the advice of the DSMB, the study would continue at the last dose of 500.10^4 cells/kg, and then be terminated (cell line exhausted).

Conditioning regimens : no restriction

The use of DLI in case of mixed chimerism or relapse is permitted after the clone infusion if necessary. In case of acute GVHD post CTL clone infusion, ganciclovir will be administered (at the dose of 5 mg/kg twice daily) for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients HLA-DPB1*04:01 positive, with confirmed diagnosis of hematologic malignancies (AML, Myelodysplasic and myeloproliferative syndrome, ALL, non-Hodgkin's lymphoma, Hodgkin's disease, CLL), undergoing an allo-HSCT using a HLA-DPB1*04:01 negative donor.
* The graft can be PBSC (peripheric blood stem cells) or bone marrow.
* Patients aged between 18-75 years.
* Patients in complete remission or >50% of response (for lymphoma) at time of transplant.
* have a donor with no contra-indications for mobilization of peripheral blood stem cells using G-CSF (colony-stimulating factors)
* Affiliation number to the National Health Care System
* Lack of reactivity of the clone against the donor's cells (PHA-blasts prepared for from PBMCs).
* For cord blood transplants: cord blood must be HLA-DPB1*04:01 negative and the HLA compatibility (A, B, DR) between the cord blood and the recipient must be 4/6, 5/6 or 6/6.
* ECOG <=2 or Karnofsky >60%
* neutrophils ≥ 1 000 cells /μl and/or platelets ≥ 50 000 cells/μl (growth factor allowed)

Exclusion Criteria:

* pregnant or breastfeeding woman
* patient refusing contraception measure
* minor
* Adult patients under guardianship, curatorship or justice protection
* Patients with post-transplant relapse within the clone injection time (before D100)
* Karnofsky performance score below 60%or ECOG >2
* Acute and chronic heart failure (NYHA Class III or IV) or symptomatic ischemic heart disease.
* Severe liver failure (bilirubin >30 µmoles/L, SGPT (Serum Glutamo-Oxalacetic Transaminase)> 4 X upper limit of normal).
* Impaired renal function (creatinine clearance < 30 ml/min)
* Acute GVHD > grade 1
* Active uncontrolled infection.
* Denied to provide informed consent
* Severe neurological or psychiatric disorders as determined by the study physician.
* Treatment with other investigational drugs following allogeneic transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
determine maximal tolerated dose of infusion of a third party suicide gene-transduced anti-HLA-DPB1*04:01 CD4+ T cell clone in HLA-DPB1*04:01 tumor positive recipients receiving an allo-HSCT from a HLA-DPB1*04:01 negative alternative donor. | 4 weeks after CTL injection
  the most likely side effects of the injection of the clone is the induction of an acute GVHD (severity measured by organ staging and overall clinical grading).
  acute GVHD will be evaluated for each patient. Maximal tolerated dose is defined as : none acute GVHD for 3 patients on 3 or for at least 5 patients on 6.
  A standard phase 1 dose-escalation study will be used:
  Level 1: 1 x 104 cells/kg of recipient, Level 2: 5 x 104 cells/kg, Level 3: 25 x 104 cells/kg, Level 4: 50 x 104 cells/kg, Level 5: 100 x 104 cells/kg After study of toxicity of the 4 injected patients, choice has been made to stop the CRM method to choose the dose and to test only 2 doses for each last patients : 100 x 10^4 cells/kg (actual level 5) and 500 x 10^4 cells/kg (choice based on compassionnal injections data at the level 5)

SECONDARY OUTCOMES:
survival and persistence of the clone injected | 6 hours after clone injection, 8 days post-injection, 15 days post-injection, 30 days post-injection, 60 days post-injection, 6 months post injection, 12 months post injection
  The survival of the clone will be tracked by PCR (polymerase chain reaction) during the 60 first days post injection as well as 6 and 12 months post injection in the blood and in the marrow
immune reconstitution | day of clone injection, 30 days after clone injection, 60 days after clone injection, 9 months after clone injection, 12 months after clone injection
  T cell reconstitution will be evaluated by measuring the levels of CD4+, CD8+, Natural Killer cells
incidence of relapse | 12 months post allograft
  Cumulative incidence of relapse
survival | 12 months post allograft
  event free survival, overall survival
GVHD incidence | 12 months post allograft
  cumulative incidence of acute and chronic GVHD
mortality | 12 months post allograft
  death not related to relapse
complete remission | 12 months post allograft
  for lymphoma patients in partial response before allograft
side effects of Clone | 12 months post allograft
  events related to clone (except GVHD)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nantes, Nantes, France